CLINICAL TRIAL: NCT02067195
Title: Aggressive Hydration in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention to Prevent Contrast-Induced Nephropathy, A Randomized, Controlled Trial REduction of riSk of Contrast-Induced Nephropathy followINg carDiac Catheterization 1
Brief Title: Aggressive hydraTion in Patients With ST -Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention to prevenT Contrast-Induced Nephropathy
Acronym: ATTEMPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Chinese PLA General Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Jiyan Chen, MD, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSC20140222
Record Dates: First submitted 2014-02-16; First posted 2014-02-20 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: acute myocardial infarction,contrast,coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guideline Hydration (Active Comparator): No hydration for patients without chronic kidney disease(CrCl<60ml/min),or Receiving hydration with a 1 mL/kg bolus of intravenous isotonic saline (0.9% sodium chloride) after diagnosis of chronic kidney disease until 24 hours after PCI. Hydration rate was reduced to 0.5 mL/kg per hour in patients with New York Heart Association class III or KillipⅡ/Ⅲ.
  Interventions: Drug: Receiving hydration with a 1 mL/kg bolus of intravenous isotonic saline (0.9% sodium chloride)
- Adequate Hydration (Active Comparator): Receiving hydration with a 3 mL/kg.hour bolus of intravenous isotonic saline (0.9% sodium chloride) from randomization to the end of the procedure, the measurement of LVEDP was conducted after the procedure, a sliding-scale hydration was employed in the LVEDP-guided hydration arm that was based on LVEDP for 2 hours: 5 ml/kg/hr for LVEDP <13 mmHg, 3 ml/kg/hr for LVEDP 13-18 mmHg, and >1.5 ml/kg/hr for LVEDP >18 mmHg, whereas,0.5 ml/kg/hr for LVEDP >20 mmHg, continue hydration with a 1 mL/kg until 24 hours after procedure. Hydration rate was reduced to 0.5 mL/kg per hour in patients with New York Heart Association class III or KillipⅡ/Ⅲ.
  Interventions: Drug: 3 mL/kg.hour bolus of intravenous isotonic saline (0.9% sodium chloride)

INTERVENTIONS:
Drug: Receiving hydration with a 1 mL/kg bolus of intravenous isotonic saline (0.9% sodium chloride) — No hydration for patients without chronic kidney disease(CrCl<60ml/min),or Receiving hydration with a 1 mL/kg bolus of intravenous isotonic saline (0.9% sodium chloride) after diagnosis of chronic kidney disease until 24 hours after PCI. Hydration rate was reduced to 0.5 mL/kg per hour in patients with New York Heart Association class III or KillipⅡ/Ⅲ.
  Other Names: Guideline Hydration
  Arms: Guideline Hydration
Drug: 3 mL/kg.hour bolus of intravenous isotonic saline (0.9% sodium chloride) — Receiving hydration with a 3 mL/kg.hour bolus of intravenous isotonic saline (0.9% sodium chloride) from randomization to the end of the procedure, the measurement of LVEDP was conducted after the procedure, a sliding-scale hydration was employed in the LVEDP-guided hydration arm that was based on LVEDP for 2 hours: 5 ml/kg/hr for LVEDP <13 mmHg, 3 ml/kg/hr for LVEDP 13-18 mmHg, and >1.5 ml/kg/hr for LVEDP >18 mmHg, whereas,0.5 ml/kg/hr for LVEDP >20 mmHg, continue hydration with a 1 mL/kg until 24 hours after procedure. Hydration rate was reduced to 0.5 mL/kg per hour in patients with New York Heart Association class III or KillipⅡ/Ⅲ.
  Other Names: Adequate Hydration
  Arms: Adequate Hydration

SUMMARY:
To compare the efficacy of 2 different hydration strategies, hydration according to clinical guideline and adequate hydration, on contrast-induced nephropathy in patients with STEMI undergoing primary PCI to investigate the possible beneficial role of periprocedural adequate hydration.

DETAILED DESCRIPTION:
all consecutive patients with STEMI，age at least 18 years, who were candidates for primary PCI at our institution were considered for enrollment in the present study. Initial exclusion criteria were contrast medium administration within the previous 14 days, end-stage renal failure requiring dialysis, and refusal to give informed consent. Eligible patients were randomly assigned in a 1:1 ratio to receive preprocedure and postprocedure hydration (adequate hydration group), hydration according to clinical guideline (guideline hydration group，control group )

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients with STEMI, age at least 18 years, who were candidates for primary PCI were considered for enrollment.

Exclusion Criteria:

* contrast medium administration within the previous 14 days or follow 72 hours,
* end-stage renal failure or renal transplantation, and refuse PCI or dead during the procedure,
* heart failure of cardiac shock or New York Heart Association class IV,
* recent acute kidney injury defined as an absolute increase of 0.5 mg/dl in serum creatinine over baseline in the past 24h
* ,the presence of lactation, pregnancy,
* malignant tumour or life expectancy less than 1 year,
* allergy to contrast, peri-procedural receipt of metformin non-steroidalanti-inflammatory drugs in the past 48h and during the study period,
* planned renal catheterization or heart valvular surgery。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Contrast-Induced Nephropathy | 72 hours
  defined as a greater than 25% or an absolute increase of 0.5 mg/dl in serum creatinine over baseline during the first 48- 72 h post-procedure
Contrast Induced Acute Kidney Injury | 24 hours
  defined as a greater than 10% or an absolute increase of 0.3mg/dl in serum Cystatin C over baseline during the first 24 h post-procedure.

SECONDARY OUTCOMES:
contrast-induced acute kidney injury | 48 hours
  defined as a greater than 50% or an absolute increase of 0.3 mg/dl in serum creatinine over baseline during the first 48h post-procedure
Composite contrast-induced acute kidney injury | 48 hours
  Defined as an absolute increase of 0.3 mg/dl in serum creatinine over baseline during the first 48h post-procedure and as a greater than 10% in Cystatin C over baseline during the first 24h post-procedure
Persistent renal damage | 3 months
  Defined as a residual impairment of renal function indicated by a reduction of creatinine clearance more than 25% at 3 months in comparison with baseline
Alteration of renal function | 72 hours
  defined as the alteration of creatinine clearance and estimated glomerular filtration rate (GFR) by using Cystatin C over baseline during the first 48- 72 h post-procedure
Severe adverse renal events | 1 year
  Including contrast-induced nephropathy requiring renal replacement therapy and death caused by contrast-induced nephropathy
Major adverse cardiovascular events | 1 year
  Major adverse cardiovascular events included death, re- current myocardial infarction, repeated urgent revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, MD, Principal Investigator — Guangdong Cardiovascular Institute,Guangdong General Hospital; Yong Liu, MD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Guo W, Song F, Chen S, Zhang L, Sun G, Liu J, Chen J, Liu Y, Tan N; RESCIND group. The relationship between hyperuricemia and contrast-induced acute kidney injury undergoing primary percutaneous coronary intervention: secondary analysis protocol for the ATTEMPT RESCIND-1 study. Trials. 2020 Jun 24;21(1):567. doi: 10.1186/s13063-020-04505-w. PMID 32580757
- [Derived] Liu J, Guo Z, Lei L, Sun G, He Y, Song F, Chen J, Tan N, Chen S, Liu Y. Statistical analysis plan for aggressive hydraTion in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention to prevenT contrast-induced nephropathy (ATTEMPT) study. Ann Transl Med. 2020 Apr;8(7):457. doi: 10.21037/atm.2020.03.192. PMID 32395501
- [Derived] Song F, Sun G, Liu J, Chen JY, He Y, Liu L, Liu Y; RESCIND group. Efficacy of post-procedural oral hydration volume on risk of contrast-induced acute kidney injury following primary percutaneous coronary intervention: study protocol for a randomized controlled trial. Trials. 2019 May 27;20(1):290. doi: 10.1186/s13063-019-3413-5. PMID 31133052
- [Derived] Liu Y, Chen JY, Huo Y, Ge JB, Xian Y, Duan CY, Chen SQ, Jiang W, Chen PY, Tan N; RESCIND group. Aggressive hydraTion in patients with ST-Elevation Myocardial infarction undergoing Primary percutaneous coronary intervention to prevenT contrast-induced nephropathy (ATTEMPT): Study design and protocol for the randomized, controlled trial, the ATTEMPT, RESCIND 1 (First study for REduction of contraSt-induCed nephropathy followINg carDiac catheterization) trial. Am Heart J. 2016 Feb;172:88-95. doi: 10.1016/j.ahj.2015.10.007. Epub 2015 Oct 20. PMID 26856220